CLINICAL TRIAL: NCT07143669
Title: A Multicenter Screening Study to Characterize the Prevalence of the KIT D816V Mutation in Patients With Suspected Clonal Mast Cell Disease
Brief Title: Screening Study for KIT D816V Mutated Mast Cell Disease in Select Populations
Status: Recruiting | Type: Observational
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-MCAD-1101
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Clonal Mast Cell Disease; KIT D816V Mutation; Suspected KITD816V Mutated Clonal Mast Cell Disease
Keywords: Mast Cell Activation Disorder; MDS/MPN Overlap Syndrome; Chronic Myelomonocytic Leukemia; Hypermobility Syndrome Disorder; Postural Orthostatic Tachycardia Syndrome; Early Onset Osteoporosis
MeSH Terms: conditions — Mastocytosis; Leukemia, Myelomonocytic, Chronic; Postural Orthostatic Tachycardia Syndrome | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Serum, Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Participants with symptoms of mast cell activation (SMAC).
  Interventions: Other: Screening
- Cohort 2: Participants with select diseases with suspected clonal mast cell involvement.
  Interventions: Other: Screening
- Cohort 3: Participants with chronic myelomonocytic leukemia or myelodysplastic syndrome/myeloproliferative neoplasm not otherwise specified.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — After providing informed consent and relevant medical history data, samples will be collected from participants with suspected clonal mast cell disease.

SUMMARY:
This is a multicenter screening study to characterize the prevalence of the KIT D816V mutation in participants with suspected clonal mast cell disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Cohort 1 participants must meet inclusion criteria for either SMAC-A or SMAC-B:

  1. SMAC-A
* Documented anaphylaxis due to Hymenoptera venom with cardiovascular symptoms or
* Documented anaphylaxis without known trigger(s) or allergen(s) warranting hospitalization, emergency room visit, and/or epinephrine with cardiovascular symptoms 2. SMAC-B
* Episodic or recurrent signs and symptoms consistent with mast cell activation without known triggers or allergens in at least 2 of the following organ systems: skin, respiratory/naso-ocular, gastrointestinal tract, or cardiovascular.
* Any clinical response on one or more optimally dosed therapies intended to mitigate mast cell mediators, as determined by the Investigator.
* Cohort 2 participants must have confirmed, known diagnosis of 1 of the following criteria:

  1. Either hypermobile Ehlers-Danlos syndrome or documented history of hypermobility spectrum disorder.
  2. Postural orthostatic tachycardia syndrome with one or more systemic symptoms.
  3. Early onset (≤50 years old) osteoporosis or osteopenia.
* Cohort 3 participants must have documented diagnosis of 1 of the following, according to World Health Organization 5th edition criteria: chronic myelomonocytic leukemia or myelodysplastic syndrome/myeloproliferative neoplasm not otherwise specified.

Key Exclusion Criteria:

* Participants previously diagnosed with any of the following:

  1. Monoclonal mast cell activation syndrome with a known KIT mutation
  2. Cutaneous mastocytosis only (that is, no documentation of systemic mast cell disease via bone marrow biopsy)
  3. Any subtype of systemic mastocytosis
  4. Mast cell sarcoma
* Cohort 2 only: Osteopenia or osteoporosis attributed to known genetic, endocrine, nutritional, or other medical conditions.

Note: Additional protocol-defined criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with suspected clonal mast cell disease
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants in Cohort 1 with KIT D816V Mutation in Peripheral Blood as Measured by Digital Droplet Polymerase Chain Reaction (ddPCR) | Day 1
Proportion of Participants in Cohort 1 with KIT D816V Mutation in Peripheral Blood as Measured by Ultra-sensitive KIT D816V by Rolling Circle Amplification (RCA) Assay | Day 1

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Kaiser Permanente San Diego, San Diego, California
  - Allergy & Asthma Clinical Research of the Bay Area, Walnut Creek, California
  - Emory University, Atlanta, Georgia
  - Midwest Allergy Sinus Asthma, Normal, Illinois
  - AllerVie Health, Glenn Dale, Maryland
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Care Access Research, Warwick, Rhode Island
  - AIR Care, Dallas, Texas